CLINICAL TRIAL: NCT06994663
Title: Evaluating the Accuracy of Commercially Available Finger Pulse Oximeters in a Hospital Setting
Brief Title: Finger Pulse Oximeters in Hosptial Setting
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 010501
Record Dates: First submitted 2018-01-17; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hypoxia; Respiratory Failure With Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulse oximetry is a well-established, non-invasive measurement tool used to estimate arterial oxygen saturation. The accuracy of these cheap, readily available finger pulse oximeters has not been robustly assessed in a clinical trial however.

It is vital for clinical practice that this technology is reliable in tracking changes in oxygen saturations at times of ill health as varying physiological parameters may, in theory, contribute to inaccurate readings.

This study will investigate whether these new devices provide a sufficiently accurate measurement of oxygen levels in the blood (when compared to arterial blood gas sampling) to endorse their use in routine hospital practice.

DETAILED DESCRIPTION:
The investigators propose to assess the margins of agreement between newer commercially available finger pulse oximeters and arterial blood gases in a hospital setting.

Eligible participants requiring blood gas assessment will be identified by members of the clinical team, who will inform the research team investigator. Arterial blood gas sampling is usually performed in patients who are breathless with low oxygen levels.

At the time of arterial blood gas sampling, the three finger pulse oximeters will be placed on each of three fingers of the participant.

The pulse oximeters are small cubic devices, each about the size of a matchbox that sits lightly over the fingernail. Light is emitted from the device and passes through the nailbed.The blood oxygen levels can then be estimated by measuring the absorption of different wavelengths of light. The participant will be asked to remain seated and still for 2mins until steady state is achieved. At this time readings will be taken from each machine.

The contemporaneous measurements of oxygen saturation using gold standard, invasive arterial blood gas sampling and new non-invasive portable pulse oximeters will allow the investigators to evaluate the accuracy of these devices and evaluate their clinical usefulness in the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Hospital inpatients deemed by the clinical team to require arterial blood gas sampling (Typically this would represent patients who are complaining of breathlessness or who have low oxygen saturations)
* Informed consent

Exclusion Criteria:

* Inability to consent (including language barrier)
* Age <16 years old

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In hospital patients requiring blood gas sampling (Typically this would represent patients who are complaining of breathlessness or who have low oxygen saturations)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Correlation | Baseline
  The handheld pulse oximeters will exhibit a good correlation as evidenced by the Intraclass correlation coefficient of 0.75. The cohort patients who were deemed by their treating physician to require an arterial blood gas sample had simultaneous SpO2 readings using 3 pulse oximeters (TempIR-Oxy, Jumper JPD-500A and Nonin Vantage 9590). Data were analysed using Pearson correlation co-efficient (r) and Bland Altman bias plot.